CLINICAL TRIAL: NCT00161330
Title: A Multicenter Randomized Controlled Trial of Antibiotic Treatment in Children With Urinary Tract Infections: Oral Amoxicillin/Clavulanic Acid vs Initial iv Ceftriaxone.
Brief Title: Oral vs Initial Intravenous Antibiotic Treatment of Urinary Tract Infections in Children: a RCT
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: University of Padova (Other)
Collaborators: Regione Veneto (Other); IL Sogno di Stefano (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRIS 1
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2020-12-14 (Actual); Status verified 2004-07

CONDITIONS: Urinary Tract Infections
Keywords: urinary tract infection,; antibiotic treatment; childhood; amoxicilline/clavulanic acid; ceftriaxone; renal ultrasonography; renal scintigraphy
MeSH Terms: conditions — Urinary Tract Infections | interventions — Amoxicillin; Clavulanic Acid; Ceftriaxone

INTERVENTIONS:
Drug: oral amoxicilline/clavulanic acid
Drug: iv ceftriaxone

SUMMARY:
The main objectives of the study are

1. to compare the efficacy of oral vs initial iv antibiotic treatment in children with a first episode of UTI
2. to assess the diagnostic power of the various imaging technique (renal ultrasonogram, voiding cystourethrogram, and renal scanning with technetium-99m-labeled dimercaptosuccinic acid)

DETAILED DESCRIPTION:
Background. Upper urinary tract infections (UTIs) are common in children, but attitudes toward the diagnosis and the acute treatment are heterogeneous among pediatricians and pediatric nephrologists. In effect the choice of antibiotic regimens is largely empirical and based on local practice, with no rationale for the choice of oral or parenteral administration. A retrospective study (1993-97) showed that in 1333 (36 % M) hospitalized children because of a prove UTI, parenteral antibiotic was given initially to 756 (57.2%) of the population studied.

We are aware of a unique randomized clinical trial, which has shown no differences in the short term (mean time to defervescence) and long term outcomes (symptomatic reinfections and renal scarring) of children receiving oral cefixime for 14 days versus vs initial iv cefotaxime for 3 days, followed by oral cefixime for 11 days.

The management of patients with UTI consists not only in antibiotic treatment of acute episodes, but also in the global evaluation of any risk factors. Current recommendations for imaging of the urinary tract are not based on prospective studies of outcomes (development of renal scars). A recent publication (Hoberman et al) suggests that renal ultrasonography and DMSA scanning at the time of acute illness are of limited value and recommends the routine use of voiding cystourethrography to identify children with reflux.

Aims.

Main objective of the study is:

1. to compare the efficacy of oral vs initial iv antibiotic treatment in children with a first episode of UTI;

Secondary objectives of the study are:

1. to assess the diagnostic power of the various imaging technique (renal ultrasonogram, voiding cystourethrogram, and renal scanning with technetium-99m-labeled dimercaptosuccinic acid);
2. to evaluate a possible role of genetic polymorphisms implicated in the evolution of kidney damage
3. to obtain area based protocols for the treatment and hospitalization of children with UTI.

Study design. A randomised, controlled, open-label, 2-armed, parallel-group study comparing the safety and efficacy of oral antibiotic (10 days of amoxicillin + clavulanic acid 50 mg/Kg/day), vs initial iv treatment (ceftriaxon 50 mg/Kg/day until defervescence) followed by oral treatment (amoxicillin + clavulanic acid) for a total of 10 days, in children with a first episode of UTI.

Criteria for the diagnosis of upper UTI upon entry

1. Urinalysis (two concordant consecutive tests)

   * Urine WBC ( higher 25/ul = 1+ with dipstick)
2. Urine culture (two concordant consecutive tests)

   * Growth of only one microorganism > 100,000 CFU
3. Fever higher than 38°C (NB: in the first 6 months of life fever is not an essential criterion)
4. Inflammation indices in the first 48 hours ESR higher than 30 and/or C-reactive Protein more than 3 times the upper limit of normal values
5. Neutrophils higher than the normal values for age

The diagnosis of upper UTI is made by presence of criteria 1, 2 and at least two of the others.

Assuming that 15% of children with pyelonephritis and treated iv will develop renal scars at the 12 month DMSA, defining efficacy as an incidence of 10% per group and setting alfa error = 0.05 and power = 80%, 220 patients per group (i.e. a total of 440 patients) are required.

The computer generated randomization list is stratified for hospital, sex and age (< o > than 2 years) and based on variable blocks of 10 or more.

Primary end points are:1. Duration of fever (>38°), 2. Sterilization of the urine, 3. Reduction of the blood inflammatory indices, 4. Incidence of renal scarring documented at 12 month.

The imaging diagnostic work-up is as follow: sonography (US) of the kidney and the bladder and DMSA renal scintigraphy within 10 days from onset of antibiotic treatment and at the end of the study (12 months), voiding cystourethrography (VC) 1-2 months after UTI.

ELIGIBILITY:
Inclusion Criteria:

* age between 2 months and 6 years,
* normal renal function
* first episode of upper UTI (fever, 2 consecutive positive urinalysis, later confirmed by 2 cultures and high blood inflammation indices)

Exclusion Criteria:

* documented previous urinary tract malformation (prenatal ultrasound)
* seriously compromised general conditions (such as sepsis or vomit)
* hypersensitivity to the antibiotics considered.

Ages: 2 Months to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 440
Dates: Start 2000-06; Study Completion 2005-07

PRIMARY OUTCOMES:
1. Duration of fever (>38°),
2. Sterilization of the urine,
3. Reduction of the blood inflammatory indices,
4. Incidence of renal scarring documented at 12 month.

CONTACTS AND LOCATIONS:
Overall Officials: Graziella Zacchello, Professor, Study Chair — Nephrology, dialysis and transplant unit, Pediatric Departement, Azienda ospdealiera-università, Padova; Antonella Toffolo, Dr, Principal Investigator — Pediatric Unit, Ospedale di Oderzo, Italy; Giovanni Montini, Dr, Principal Investigator — Nephrology, Dialysis and Transplant Unit, Pediatric Departement, Azienda Ospedaliera - Università, Padova Italy

REFERENCES:
- [Background] Ghiro L, Cracco AT, Sartor M, Comacchio S, Zacchello G, Dall'Amico R; Veneto Urinary Tract Infection Study Group. Retrospective study of children with acute pyelonephritis. Evaluation of bacterial etiology, antimicrobial susceptibility, drug management and imaging studies. Nephron. 2002 Jan;90(1):8-15. doi: 10.1159/000046308. PMID 11744799
- [Background] Hoberman A, Wald ER, Hickey RW, Baskin M, Charron M, Majd M, Kearney DH, Reynolds EA, Ruley J, Janosky JE. Oral versus initial intravenous therapy for urinary tract infections in young febrile children. Pediatrics. 1999 Jul;104(1 Pt 1):79-86. doi: 10.1542/peds.104.1.79. PMID 10390264
- [Background] Downs SM. Technical report: urinary tract infections in febrile infants and young children. The Urinary Tract Subcommittee of the American Academy of Pediatrics Committee on Quality Improvement. Pediatrics. 1999 Apr;103(4):e54. doi: 10.1542/peds.103.4.e54. PMID 10103346
- [Background] Jakobsson B, Esbjorner E, Hansson S. Minimum incidence and diagnostic rate of first urinary tract infection. Pediatrics. 1999 Aug;104(2 Pt 1):222-6. doi: 10.1542/peds.104.2.222. PMID 10428998
- [Background] Cornu C, Cochat P, Collet JP, Delair S, Haugh MC, Rolland C. Survey of the attitudes to management of acute pyelonephritis in children. GEP. Pediatr Nephrol. 1994 Jun;8(3):275-7. doi: 10.1007/BF00866331. PMID 7917849
- [Background] Jodal U. Treatment trials on children with acute pyelonephritis. Pediatr Nephrol. 1994 Jun;8(3):278-9. doi: 10.1007/BF00866332. No abstract available. PMID 7917850
- [Background] Hoberman A, Charron M, Hickey RW, Baskin M, Kearney DH, Wald ER. Imaging studies after a first febrile urinary tract infection in young children. N Engl J Med. 2003 Jan 16;348(3):195-202. doi: 10.1056/NEJMoa021698. PMID 12529459
- [Background] Levtchenko EN, Ham HR, Levy J, Piepsz A. Attitude of Belgian pediatricians toward strategy in acute pyelonephritis. Pediatr Nephrol. 2001 Feb;16(2):113-5. doi: 10.1007/s004670000531. PMID 11261676
- [Derived] Hewitt IK, Zucchetta P, Rigon L, Maschio F, Molinari PP, Tomasi L, Toffolo A, Pavanello L, Crivellaro C, Bellato S, Montini G. Early treatment of acute pyelonephritis in children fails to reduce renal scarring: data from the Italian Renal Infection Study Trials. Pediatrics. 2008 Sep;122(3):486-90. doi: 10.1542/peds.2007-2894. PMID 18762516
- [Derived] Montini G, Toffolo A, Zucchetta P, Dall'Amico R, Gobber D, Calderan A, Maschio F, Pavanello L, Molinari PP, Scorrano D, Zanchetta S, Cassar W, Brisotto P, Corsini A, Sartori S, Da Dalt L, Murer L, Zacchello G. Antibiotic treatment for pyelonephritis in children: multicentre randomised controlled non-inferiority trial. BMJ. 2007 Aug 25;335(7616):386. doi: 10.1136/bmj.39244.692442.55. Epub 2007 Jul 4. PMID 17611232